CLINICAL TRIAL: NCT04592068
Title: Deep Learning-Based Automated Classification of Multi-Retinal Disease From Fundus Photography
Brief Title: AI Classifies Multi-Retinal Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Tulip Partner Technology Co., Ltd, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: Retinal multi diseases
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-10

CONDITIONS: Deep Learning; Retinal Diseases
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retinal multi-diseases diagnosed by DL algorithm
  Interventions: Device: Retinal multi-diseases diagnosed by DL algorithm
- Retinal multi-diseases diagnosed by expert panel
  Interventions: Other: Retinal multi-diseases diagnosed by expert panel

INTERVENTIONS:
Device: Retinal multi-diseases diagnosed by DL algorithm — DL algorithm automatically classify multi-diseases from fundus photography and differentiate major vision-threatening conditions and other retinal abnormalities.
  Groups: Retinal multi-diseases diagnosed by DL algorithm
Other: Retinal multi-diseases diagnosed by expert panel — Expert panel classifies multi-diseases from fundus photography and differentiate major vision-threatening conditions and other retinal abnormalities.
  Groups: Retinal multi-diseases diagnosed by expert panel

SUMMARY:
The objective of this study is to establish deep learning (DL) algorithm to automatically classify multi-diseases from fundus photography and differentiate major vision-threatening conditions and other retinal abnormalities. The effectiveness and accuracy of the established algorithm will be evaluated in community derived dataset.

DETAILED DESCRIPTION:
Retinal diseases seriously threaten vision and quality of life, but they often develop insidiously. To date, deep learning (DL) algorithms have shown high prospects in biomedical science, particularly in the diagnosis of ocular diseases, such as diabetic retinopathy, age-related macular degeneration, retinopathy of prematurity, glaucoma, and papilledema. However, there is still a lack of a single algorithm that can classify multi-diseases from fundus photography.

This cross-sectional study will establish a DL algorithm to automatically classify multi-diseases from fundus photography and differentiate major vision-threatening conditions and other retinal abnormalities. We will use the receiver operating characteristic (ROC) curve to examine the ability of recognition and classification of diseases. Taken the results of the expert panel as the gold standard, we will use the evaluation indexes, such as sensitivity, specificity, accuracy, positive predictive value, negative predictive value, etc, to compare the diagnostic capacity between the AI recognition system and human ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* fundus photography around 45° field which covers optic disc and macula
* complete patient identification information;

Exclusion Criteria:

* incomplete patient identification information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community derived dataset
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Area under curve | 1 week
  We will use the receiver operating characteristic (ROC) curve to examine the ability of recognition and classification of diseases. Taken the results of the expert panel as the gold standard, we will use the area under curve to compare the diagnostic capacity between the AI recognition system and human ophthalmologist.
Sensitivity and specificity | 1 week
  Taken the results of the expert panel as the gold standard, we will use sensitivity and specificity to compare the diagnostic capacity between the AI recognition system and human ophthalmologist.
Positive and negative predictive value | 1 week
  Taken the results of the expert panel as the gold standard, we will use positive and negative predictive value to compare the diagnostic capacity between the AI recognition system and human ophthalmologist.
Accuracy | 1 week
  Taken the results of the expert panel as the gold standard, we will use accuracy to compare the diagnostic capacity between the AI recognition system and human ophthalmologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-Bin Wei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gu C, Wang Y, Jiang Y, Xu F, Wang S, Liu R, Yuan W, Abudureyimu N, Wang Y, Lu Y, Li X, Wu T, Dong L, Chen Y, Wang B, Zhang Y, Wei WB, Qiu Q, Zheng Z, Liu D, Chen J. Application of artificial intelligence system for screening multiple fundus diseases in Chinese primary healthcare settings: a real-world, multicentre and cross-sectional study of 4795 cases. Br J Ophthalmol. 2024 Feb 21;108(3):424-431. doi: 10.1136/bjo-2022-322940. PMID 36878715